CLINICAL TRIAL: NCT01468545
Title: Prospective, Non-interventional, Multi-centre Study. The Observation Period for Each Subject Covers 1 Year of Treatment. One Initial Visit and 4 Follow-up Visits Every 3 Months and One Extra Educational Reinforcement at Baseline and at 6 Months Will be Given to a Group of Patients.
Brief Title: Educational Training Influence in Patients With PAH(Pulmonary Artery Hypertension) on Inhaled Ventavis Treatment Adherence Evaluated Trough INSIGHT System
Acronym: Inventa
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Dra. Pilar Escribano Subías - Coordinator - HU 12 de Octubre - Madrid (Spain) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 15554; BAY-ILO-2010-01 (Other: company internal)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Education; Ventavis; Adherence; PAH; Pulmonary artery hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension | interventions — Iloprost

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Other: Iloprost (Ventavis inhaled, BAYQ6256)
- Group 2
  Interventions: Other: Iloprost (Ventavis inhaled, BAYQ6256)

INTERVENTIONS:
Other: Iloprost (Ventavis inhaled, BAYQ6256) — An extra educational reinforcement at baseline and at 6 months will be given to a group of patients
  Groups: Group 1
Other: Iloprost (Ventavis inhaled, BAYQ6256) — No extra educational reinforcement.
  Groups: Group 2

SUMMARY:
Ventavis it's a treatment for pulmonary hypertension, administered by an inhaler called I-Neb.

In these patients, the non compliance of the treatment becomes its ineffective and increases the complications and mortality of the disease.

It is therefore important to know which the adherence of patients to their treatment is and try to promote it.

One possibility to reach a good level of adherence is the patient education regarding the drug administration and also to comply as better is possible the recommendations of the physician.

For this reason, the objective of our study is to demonstrate improvement in the level of treatment compliance when they follow a strategy of continuing education, assessed by the device and software called Insight.

The only special procedure to participate in the study then is that patients involved could receive more training than usual.

Investigators expect involving in this study around 50 patients in treatment with Ventavis and diagnosed of Pulmonary Arterial Hypertension in 10-12 hospitals throughout Spain.

The patients who participated in the study will be followed for 12 months from inclusion in the study and will perform around 5 visits in total.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years of age.
* Patients in New York Heart Association (NYHA) functional class II-IV pulmonary hypertension who are treated with Ventavis at least three months before and who use -neb ® AAD ® system.
* Patients who accepted participation in the study and sign informed consent.
* Patients with ability to understand and follow the instructions and are able to participate for the duration of the study.

exclusion Criteria:

* Patients with severe cognitive impairment.
* Geographically unstable patients who can not be followed during the 12 month study.
* Patients who have a life expectancy of at least 12 months.
* Patients who are participating in another study at the time of inclusion. .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 PAH patients in treatment with Ventavis.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The influence of educational training on Ventavis treatment compliance through the Insight system | 12 months

SECONDARY OUTCOMES:
Number of events requiring non-planned visit or hospital admission related to PAH(Pulmonary Artery Hypertension), depending on the education sessions received. | 12 months
Number of events due to Inhaler-related errors | 12 months
The difference of adherence patient information (subjective data) through the Morisky-Green questionnaire and the one shown by the Insight registry (objective data) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Spain